CLINICAL TRIAL: NCT02732015
Title: Effects of Rolapitant on Nausea/Vomiting in Patients With Sarcoma Receiving Multi-Day Highly Emetogenic Chemotherapy (HEC) With Doxorubicin and Ifosfamide Regimen (AI)
Brief Title: Rolapitant Hydrochloride in Preventing Nausea/Vomiting in Patients With Sarcoma Receiving Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated per PI's request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-0587; NCI-2016-00801 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0587 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-04-04; First posted 2016-04-08 (Estimated); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced Sarcoma
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; fosaprepitant; Aprepitant; Ifosfamide; Mesna; Ondansetron; rolapitant; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (rolapitant hydrochloride) (Experimental): Patients receive treatment as in part I. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  CHEMOTHERAPY: All patients receive doxorubicin IV over 72 hours, mesna IV, and ifosfamide IV over 3 hours on days 1-4 or 1-5. Patients with sarcomas of small cell histology receive vincristine sulfate IV on day 1. Cycles repeat every 3 weeks following blood count and patient recovery from any acute toxicities.
  Interventions: Drug: Dexamethasone; Drug: Doxorubicin; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Mesna; Drug: Ondansetron; Other: Questionnaire Administration; Drug: Rolapitant Hydrochloride; Drug: Vincristine Sulfate
- Arm II (fosaprepitant dimeglumine) (Active Comparator): Patients receive dexamethasone IV and ondansetron IV on days 1-5, and fosaprepitant dimeglumine IV over 30 minutes on days 1 of cycle 2. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.
  CHEMOTHERAPY: All patients receive doxorubicin IV over 72 hours, mesna IV, and ifosfamide IV over 3 hours on days 1-4 or 1-5. Patients with sarcomas of small cell histology receive vincristine sulfate IV on day 1. Cycles repeat every 3 weeks following blood count and patient recovery from any acute toxicities.
  Interventions: Drug: Dexamethasone; Drug: Doxorubicin; Drug: Fosaprepitant Dimeglumine; Drug: Ifosfamide; Other: Laboratory Biomarker Analysis; Drug: Mesna; Drug: Ondansetron; Other: Questionnaire Administration; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Dexamethasone — Given IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxydaunomycin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Fosaprepitant Dimeglumine — Given IV
  Other Names: Emend for Injection; L-785,298; MK-0517
  Arms: Arm II (fosaprepitant dimeglumine)
Drug: Ifosfamide — Given IV
  Other Names: Asta Z 4942; Asta Z-4942; Cyfos; Holoxan; Holoxane; Ifex; IFO; IFO-Cell; Ifolem; Ifomida; Ifomide; Ifosfamidum; Ifoxan; IFX; Iphosphamid; Iphosphamide; Iso-Endoxan; Isoendoxan; Isophosphamide; Mitoxana; MJF 9325; MJF-9325; Naxamide; Seromida; Tronoxal; Z 4942; Z-4942
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mesna — Given IV
  Other Names: 2-Mercaptoethanesulfonate, Sodium Salt; Ausobronc; D-7093; Filesna; Mercaptoethane Sulfonate; Mercaptoethanesulfonate; Mesnex; Mesnil; Mesnum; Mexan; Mistabron; Mistabronco; Mitexan; Mucofluid; Mucolene; UCB 3983; Uromitexan; Ziken
Drug: Ondansetron — Given IV
  Other Names: Zofran ODT; Zuplenz
Other: Questionnaire Administration — Ancillary studies
Drug: Rolapitant Hydrochloride — Given PO
  Other Names: Rolapitant HCl; Rolapitant Hydrochloride Monohydrate; Rolapitant Monohydrochloride Monohydrate; SCH-619734; SCH619734; Varubi
  Arms: Arm I (rolapitant hydrochloride)
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized phase II trial studies how well rolapitant hydrochloride works in preventing nausea/vomiting in patients with sarcoma receiving chemotherapy. Antiemetic drugs, such as rolapitant hydrochloride, may help control or prevent nausea and vomiting in patients treated with chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the effect of rolapitant hydrochloride (rolapitant) on nausea/vomiting in patients with sarcoma receiving multi-day highly emetogenic chemotherapy (HEC) regimen of doxorubicin and ifosfamide (AI).

SECONDARY OBJECTIVES:

I. To evaluate the toxicity of rolapitant in patients receiving AI regimen. II. To evaluate the effects of rolapitant on patient reported outcomes.

OUTLINE:

PART I: Patients receive dexamethasone intravenously (IV) daily and ondansetron IV on days 1-5, and rolapitant hydrochloride orally (PO) on day 1.

PART II: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive treatment as in part I. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive dexamethasone IV and ondansetron IV on days 1-5, and fosaprepitant dimeglumine IV over 30 minutes on days 1 of cycle 2. Treatment repeats every 21 days for 6 cycles in the absence of disease progression or unacceptable toxicity.

CHEMOTHERAPY: All patients receive doxorubicin IV over 72 hours, mesna IV, and ifosfamide IV over 3 hours on days 1-4 or 1-5. Patients with sarcomas of small cell histology receive vincristine sulfate IV on day 1. Cycles repeat every 3 weeks following blood count and patient recovery from any acute toxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sarcoma which is locally advanced, at high risk for relapse or metastatic for whom treatment with doxorubicin plus ifosfamide (AI) or AI and vincristine (VAI) is indicated
* Patient must have an estimated life expectancy >= 4 months in the opinion of the investigators
* Male and females of child bearing potential must use acceptable methods of birth control which include oral contraceptives, spermicide with either a condom, diaphragm or cervical cap, use of an intrauterine device (IUD) or abstinence

  * Female patients must have a negative pregnancy test at screening
  * Female patients of childbearing potential must agree to use an acceptable method of birth control (excluding hormonal birth control methods) for 72 hours prior to admission and to continue its use during the study and for at least 30 days after the final dose
  * Male patients must agree to use an acceptable form of birth control from study day 1 through at least 30 days after the final dose
* Absolute neutrophil count (ANC) > 1500/mm^3
* Platelet count > 100,000/mm^3
* Serum creatinine < 1.5 mg/dL
* Serum bilirubin count < 1.5 x upper limit normal (ULN)
* Serum glutamic-oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) < 2.5 x ULN; for subjects with known liver metastases < 5 x ULN
* Karnofsky performance status > 60%
* Signed informed consent form
* Patients are required to read and understand English to comply with protocol requirements

Exclusion Criteria:

* Any current treatment, medical history, or uncontrolled condition, other than malignancy, (e.g., alcoholism or signs of alcohol abuse, seizure disorder, medical or psychiatric condition) that, in the opinion of the investigator, would confound the results of the study or pose any unwarranted risk in administering study drug to the subject
* Patient has a known hypersensitivity to the administration of any prescribed oral or intravenous study medication or metabolite, including but not limited to, a history of hypersensitivity to the drugs or their components, severe renal impairment, severe bone marrow suppression, or systemic infection
* Patient is a woman with a positive urine or serum pregnancy test within 3 days prior to study drug administration, is breast-feeding, or is planning to conceive children within the projected duration of the study treatment
* Patient has taken the anti-emetic agents within the last 48 hours prior to the start of treatment with study drug:

  * 5-hydroxytryptamine (HT)3 antagonists (ondansetron, granisetron, dolasetron, tropisetron, etc.); palonosetron is not permitted within 7 days prior to administration of investigational product
  * Phenothiazines (prochlorperazine, fluphenazine, perphenazine, thiethylperazine, chlorpromazine, etc.)
  * Benzamides (metoclopramide, alizapride, etc.)
  * Domperidone
  * Cannabinoids
  * Neurokinin (NK)1 antagonist (aprepitant)
  * Benzodiazepines (lorazepam, alprazolam, etc)
  * Herbal medications or preparations in doses designed to ameliorate nausea or emesis
* Patient has received systemic corticosteroids or sedative antihistamines (dimenhydrinate, diphenhydramine, etc.) within 72 hours of day 1 of the study except as premedication for chemotherapy (e.g., taxanes); subjects who are receiving inhaled steroids for respiratory conditions or topical steroids for skin disorders can be enrolled
* Patient has symptomatic primary or metastatic central nervous system (CNS) disease
* Patient has ongoing vomiting, retching, dry heaves, or clinically significant nausea caused by any etiology, or has had such symptoms within 24 hours prior to the start of day 1 of the study intervention, or has a history of anticipatory nausea and vomiting
* Patient must not have been dosed with test drug or blinded study drug in another investigational study within 30 days or 5 half-lives of the biologic activity of the test drug, whichever is longer, before the time of first study dose
* Patient who is participating in any investigational agent that is not Food and Drug Administration (FDA)-approved
* Patient has uncontrolled angina, congestive heart failure (New York Heart Association > class II or known ejection fraction < 40%), uncontrolled cardiac arrhythmia or hypertension, or acute myocardial infarction within 3 months
* Prior surgery or radiotherapy (RT) within 2 weeks of study entry
* Psychological, social, familial, or geographical reasons that would prevent scheduled visits and follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saroj Vadhan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 37 participants were consented, 1 screen failure. protocol terminated early only part I of the protocol was completed.
Groups:
- Cohort 1: Dexamethasone IV daily for 5 days (12 mg on day 1 and 8 mg on days 2-5), Ondansetron (5HT3 receptor antagonist) 16 mg IV daily for 5 days as standard of care, and Rolapitant, 180 mg was administered PO on Day 1.
- Cohort 2: Dexamethasone IV daily for 5 days (12 mg on days 1-5 ), Ondansetron (5HT3 receptor antagonist) 16 mg IV daily for 5 days as standard of care, and Rolapitant, 180 mg was administered PO on Day 1
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 9 | 27
Completed | 9 | 26
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - 8mg Dexamethasone: Dexamethasone IV daily for 5 days (12 mg on day 1 and 8 mg on days 2-5), Ondansetron (5HT3 receptor antagonist) 16 mg IV daily for 5 days as standard of care, and Rolapitant, 180 mg was administered PO on Day 1.
- Cohort 2- 12mg Dexamethasone: Dexamethasone IV daily for 5 days (12 mg on days 1-5 ), Ondansetron (5HT3 receptor antagonist) 16 mg IV daily for 5 days as standard of care, and Rolapitant, 180 mg was administered PO on Day 1
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 8mg Dexamethasone | Cohort 2- 12mg Dexamethasone | Total
Number analyzed (Participants) | 9 | 27 | 36
Age, Continuous [Median (Full Range); unit: years] | 39 [24 to 60] | 38 [19 to 59] | 38 [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 17 | 20
  Male | 6 | 10 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 27 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR) of Rolapitant Hydrochloride Administered as a Single-dose
Description: Complete response (CR) no emetic episodes and no rescue medications.
Time Frame: Days 1-10
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 9 | 26
Participants | 0 | 5

ADVERSE EVENTS:
Time Frame: collected from the time of informed consent to 30 days after last study drug administration, up to 10 days
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/26
Serious Adverse Events (participants affected / at risk) | 7/9 | 13/26
Other Adverse Events (participants affected / at risk) | 7/9 | 6/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=9) | Cohort 2 (N=26)
Neutropenic Fever (Infections and infestations) | 7 | 13
Anemia (Blood and lymphatic system disorders) | 0 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 8
Mucositis (Gastrointestinal disorders) | 5 | 5
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 | 0 (0)
Electrolytes imbalance (Skin and subcutaneous tissue disorders) | 0 | 3
Dizziness (Nervous system disorders) | 1 | 2
Throat pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Chest pain (Cardiac disorders) | 0 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 2
Uncontrolled pain (General disorders) | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chest tightness (Cardiac disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rapid heart rate (Cardiac disorders) | 0 | 1
Rectal tear (Gastrointestinal disorders) | 1 | 0
Renal insufficiency (Renal and urinary disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=9) | Cohort 2 (N=26)
Constipation (Gastrointestinal disorders) | 3 | 5
Fatigue (General disorders) | 7 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 4
Headache (Nervous system disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT02732015/Prot_SAP_000.pdf